CLINICAL TRIAL: NCT00317785
Title: A Phase II Trial of Total Body Irradiation Plus Metabolism-Based Cyclophosphamide Dosing as Preparative Therapy for Allogeneic Hematopoietic Cell Transplant for Patients With Hematological Malignancy
Brief Title: Total-Body Irradiation and Cyclophosphamide in Treating Patients Who Are Undergoing Donor Stem Cell Transplant for Hematologic Cancer and Other Diseases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 1998.00; FHCRC-1998.00; CDR0000471840 (Registry Identifier: PDQ)
Record Dates: First submitted 2006-04-24; First posted 2006-04-25 (Estimated); Last update posted 2010-05-07 (Estimated); Status verified 2010-05

CONDITIONS: Leukemia; Lymphoma; Myelodysplastic Syndromes
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; blastic phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; de novo myelodysplastic syndromes; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; previously treated myelodysplastic syndromes; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult Burkitt lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent small lymphocytic lymphoma; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; splenic marginal zone lymphoma; stage III adult Burkitt lymphoma; stage III adult Hodgkin lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Myelodysplastic Syndromes; Congenital Abnormalities; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Lymphoma, B-Cell, Marginal Zone; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cyclophosphamide; Cyclosporine; Methotrexate; Mycophenolic Acid; Sirolimus; Tacrolimus; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation

INTERVENTIONS:
Drug: cyclophosphamide
Drug: cyclosporine
Drug: methotrexate
Drug: mycophenolate mofetil
Drug: sirolimus
Drug: tacrolimus
Other: pharmacological study
Procedure: allogeneic bone marrow transplantation
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: total-body irradiation

SUMMARY:
RATIONALE: Giving total-body irradiation and chemotherapy, such as cyclophosphamide, before a donor stem cell transplant helps stop the patient's immune system from rejecting the donor's stem cells and helps stop the growth of cancer or abnormal cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving immunosuppressive therapy before or after transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well giving total-body irradiation together with cyclophosphamide works in treating patients who are undergoing donor stem cell transplant for hematologic cancer and other diseases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the potential efficacy of targeting cyclophosphamide to a metabolic endpoint when given together with total-body irradiation, in terms of day 200 nonrelapse mortality, in patients with hematologic cancer and other diseases who are undergoing allogeneic hematopoietic stem cell transplantation.

Secondary

* Determine the overall survival of patients treated with this regimen.
* Determine the rate of relapse in patients treated with this regimen.
* Determine the occurrence of sinusoidal obstruction syndrome in patients treated with this regimen.
* Determine the occurrence of acute renal failure in these patients.
* Determine the occurrence of respiratory failure in these patients.

OUTLINE:

* Conditioning regimen: Patients undergo total-body irradiation twice daily on days -6 to -4. Patients also receive cyclophosphamide IV over 1 hour on day -3 and then IV at a metabolism-based dose* on day -2.

NOTE: *Patients undergo frequent blood sampling after completion of the first cyclophosphamide infusion for pharmacokinetic studies in order to determine the dose for the second cyclophosphamide infusion.

* Allogeneic stem cell transplantation: Patients undergo allogeneic bone marrow or peripheral blood stem cell transplantation on day 0.
* Graft-versus-host disease (GVHD) prophylaxis: Patients receive GVHD prophylaxis as per the attending physician, including one of the following regimens: cyclosporine and methotrexate; tacrolimus and methotrexate; tacrolimus and mycophenolate mofetil; or sirolimus, tacrolimus, and methotrexate (as per the GVHD prophylaxis regimen chosen for each patient).

After completion of study treatment, patients are followed periodically for at least 200 days.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of a hematologic cancer or other disease that is unlikely to respond to conventional treatment, including any of the following:

  * Chronic myelogenous leukemia
  * Acute myeloid leukemia
  * Acute lymphocytic leukemia
  * Myelodysplastic syndromes
  * Lymphoma
* Patients who have bulky tumor mass must not require additional involved-field irradiation
* Planning to undergo conditioning for transplantation at the Seattle Cancer Care Alliance and University of Washington Medical Center
* Must have an HLA-matched donor available

  * No donors who are mismatched for > 1 HLA class I antigen or allele
  * Negative anti-donor lymphocytotoxic crossmatch

PATIENT CHARACTERISTICS:

* Life expectancy must not be severely limited by diseases other than malignancy
* No moribund patients
* Creatinine ≤ 1.2 mg/dL
* Oxygen saturation on room air ≥ 93%
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No HIV positivity
* No cirrhosis
* No hepatic fibrosis with bridging
* No fulminant hepatic failure
* No acute liver injury
* No persistent cholestasis
* No infection requiring systemic antibiotic or antifungal therapy
* No coronary artery disease
* No congestive heart failure requiring therapy

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior hematopoietic stem cell transplantation
* No prior radiation therapy to the liver or adjacent organs
* More than 30 days since prior cytoreductive chemotherapy for patients with a large body burden of tumor cells
* No concurrent enrollment in a phase I study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-05; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Non-relapse mortality (NRM) at 200 days

SECONDARY OUTCOMES:
Overall survival
Relapse rate
Sinusoidal obstruction syndrome (SOS)
Acute renal failure
Respiratory failure
Cause of death

CONTACTS AND LOCATIONS:
Overall Officials: George B. McDonald, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (2):
- United States (2):
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington